CLINICAL TRIAL: NCT00432198
Title: Zolpidem Postmarketing Clinical Study: A Double Blind, Placebo Controlled Group Comparative Trial in the Adolescent Patients With Insomnia
Brief Title: Zolpidem Postmarketing Study in Adolescent Patients With Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6199-JC-0001
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Insomnia
Keywords: Insomnia; Zolpidem; Adolescent
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Oral
  Interventions: Drug: Zolpidem (Myslee®)
- 2 (Experimental): Oral
  Interventions: Drug: Zolpidem (Myslee®)
- 3 (Placebo Comparator): Oral
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Zolpidem (Myslee®) — Oral
  Other Names: Myslee; FK199B
  Arms: 1; 2
Drug: placebo — Oral
  Arms: 3

SUMMARY:
To investigate the efficacy and safety of zolpidem for pediatric insomniacs in a randomized double blind-controlled trial

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as having nonorganic insomnia of nonorganic sleep disorder in ICD10
* patients whose age at the time of obtaining consent is 12 years or over and 18 years or below

Exclusion Criteria:

* patients with schizophrenia or manic-depressive illness
* patients with insomnia caused by physical diseases
* patients having a history of hypersensitivity to zolpidem
* patients with attention-deficit hyperactivity disorder

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2007-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Mean daily sleep latency for double-blind period | 2 Weeks

SECONDARY OUTCOMES:
Mean daily total hours of sleep | 2 Weeks
Mean daily frequency of intermediate awaking | 2 Weeks
Mean daily time of intermediate awaking | 2 Weeks
Impression of patient for double-blind period | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kansai Region
  - Kanto Region
  - Kyushyu Region
  - Shikoku Region

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=140